CLINICAL TRIAL: NCT01241409
Title: Pivotal Study to Assess the Bioequivalence of the To-be-Marketed Sprinkle Capsule Formulation and the Phase 3 Sprinkle Capsule Formulation of Rabeprazole Sodium in Fasted Condition and to Assess the Effect of Food on the To-be-Marketed Formulation in Healthy Adult Subjects
Brief Title: A Bioequivalence Study of 2 Formulations of Rabeprazole Sodium and Evaluation of the Effect of Food on Rabeprazole Sodium in Healthy Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: CR014830; RABGRD1007 (Other: Johnson & Johnson Pharmaceutical Research & Development, L.L.C.)
Record Dates: First submitted 2010-10-21; First posted 2010-11-16 (Estimated); Last update posted 2012-10-30 (Estimated); Status verified 2012-10

CONDITIONS: Healthy
Keywords: Healthy; Sprinkle Capsule Formulation; Rabeprazole sodium; Pharmacokinetics; Bioequivalence; Safety

ARMS (6):
- Treatment sequence ABC (Experimental)
  Interventions: Drug: Rabeprazole sodium: Treatment A; Drug: Rabeprazole sodium: Treatment B; Drug: Rabeprazole sodium: Treatment C
- Treatment sequence ACB (Experimental)
  Interventions: Drug: Rabeprazole sodium: Treatment A; Drug: Rabeprazole sodium: Treatment B; Drug: Rabeprazole sodium: Treatment C
- Treatment sequence BAC (Experimental)
  Interventions: Drug: Rabeprazole sodium: Treatment A; Drug: Rabeprazole sodium: Treatment B; Drug: Rabeprazole sodium: Treatment C
- Treatment sequence BCA (Experimental)
  Interventions: Drug: Rabeprazole sodium: Treatment A; Drug: Rabeprazole sodium: Treatment B; Drug: Rabeprazole sodium: Treatment C
- Treatment sequence CAB (Experimental)
  Interventions: Drug: Rabeprazole sodium: Treatment A; Drug: Rabeprazole sodium: Treatment B; Drug: Rabeprazole sodium: Treatment C
- Treatment sequence CBA (Experimental)
  Interventions: Drug: Rabeprazole sodium: Treatment A; Drug: Rabeprazole sodium: Treatment B; Drug: Rabeprazole sodium: Treatment C

INTERVENTIONS:
Drug: Rabeprazole sodium: Treatment A — One single oral dose of 10 mg (1 x 10-mg capsule) rabeprazole to be-marketed sprinkle capsule granule formulation administered in fasted state. After the capsules are opened, the granules will be sprinkled on applesauce (1 tablespoon).
Drug: Rabeprazole sodium: Treatment B — One single oral dose of 10 mg (2 x 5-mg capsules) rabeprazole Phase 3 sprinkle capsule granule formulation administered in fasted state. After the capsules are opened, the granules will be sprinkled on applesauce (1 tablespoon).
Drug: Rabeprazole sodium: Treatment C — One single oral dose of 10 mg (1 x 10-mg capsule) rabeprazole to be-marketed sprinkle capsule granule formulation administered after consumption of a standardized high-fat high-caloric breakfast. After the capsules are opened, the granules will be sprinkled on applesauce (1 tablespoon).

SUMMARY:
The purpose of the study is to evaluate and compare the pharmacokinetics (blood levels) of 2 sprinkle capsule formulations of rabeprazole sodium when administered without food to healthy volunteers. In addition, the pharmacokinetics of 1 formulation of rabeprazole sodium will be evaluated when administered with food to healthy volunteers.

DETAILED DESCRIPTION:
This is a randomized (study drug assigned by chance), open-label (the volunteer will know the treatment/drug they are taking), single-dose study of 2 formulations of rabeprazole sodium in healthy adult volunteers. Rabeprazole sodium is a drug used to treat patients with Gastroesophageal Reflux Disease (GERD), a condition where the esophagus (tube from throat to stomach) becomes irritated or inflamed as a result of acid that backs up into the esophagus from the stomach. All volunteers will receive 3 doses of study drug; each dose of study drug will be separated by at least 7 days. Blood samples will be collected from volunteers during the study to measure the concentration of study drug. Approximately 78 healthy volunteers will be enrolled and will participate in the study for a total of approximately 39 days. During the study, the healthy volunteer will make a total of approximately 4 visits to the study center. The 4 visits will include an initial screening visit and 3 visits to receive study drug. Volunteers will be required to stay at the study center for at least 12 hours before study drug administration and up to approximately 24 hours after study drug administration to have study procedures performed and blood samples collected to measure the concentrations of rabeprazole and its thioether metabolite (a substance produced when rabeprazole is metabolized in the body) in the plasma (ie, the clear liquid portion of blood). Volunteers will be monitored for safety throughout the study. Healthy volunteers will receive a single dose of study drug in 3 treatment periods. In each treatment period, healthy volunteers will receive one 10 mg capsule of rabeprazole sodium or two 5 mg capsules of rabeprazole sodium. The contents of study drug capsules will be sprinkled on 1 tablespoon of applesauce and administered orally (by mouth) to healthy volunteers in the morning who have fasted (not eaten) overnight and to those who have eaten a standardized breakfast.

ELIGIBILITY:
Inclusion Criteria:

* Have a body mass index (BMI) between 18 and 30 kg/m² (inclusive), and body weight not less than 50 kg
* Women must be postmenopausal (no spontaneous menses for at least 2 years), surgically sterile, abstinent, or, if of childbearing potential and sexually active, be practicing an effective method of birth control before entry and throughout the study
* Women must have a negative serum beta-human chorionic gonadotropin (hCG) pregnancy test at screening and a negative urine pregnancy test on Day -1 of each treatment period
* Men must agree to use an adequate contraception method as deemed appropriate by the investigator
* Have normal blood pressure between 90 and 140 mmHg systolic and <=90 mmHg diastolic
* Exclusion Criteria:
* Currently have, or have a history of medical illness considered by the Investigator to be clinically significant or any other illness that the investigator considers should exclude the volunteer or that could interfere with the interpretation of the study results
* Have clinically significant abnormal values for hematology, clinical chemistry or urinalysis at screening as deemed appropriate by the investigator
* Have clinically significant abnormal physical examination, vital signs or 12 lead electrocardiogram (ECG) at screening as deemed appropriate by the investigator
* Have a history of drug or alcohol abuse within the past 1 year
* Have a history of smoking or use of nicotine-containing substances within the previous 2 months
* Have had major or traumatic surgery within 12 weeks before screening or preplanned surgery or procedures that would interfere with the conduct of the study
* Known allergy to the study drug or any of the excipients of the formulation
* Known allergy to heparin or history of heparin-induced thrombocytopenia
* Use of any concomitant therapy which are drug metabolizing enzyme (cytochrome P450) inducers or inhibitors within 6 weeks before study entry and during the entire study
* Use of any prescription or nonprescription medication (including vitamins and herbal supplements), except for paracetamol, hormonal contraceptives and hormonal replacement therapy, within 14 days before the first dose of the study drug is scheduled

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 78 (Actual)
Dates: Start 2010-10; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Plasma concentrations of rabeprazole sodium | Up to 16 hours after each study drug administration
Plasma concentrations of thioether metabolite | Up to 16 hours after each study drug administration

SECONDARY OUTCOMES:
The number of participants with adverse events as a measure of safety and tolerability | Up to approximately 39 days

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- [Derived] Thyssen A, Solanki B, Gonzalez M, Leitz G, Treem W, Mannaert E. Pharmacokinetics of rabeprazole granules versus tablets, and the effect of food on the pharmacokinetics of rabeprazole granules in healthy adults-cross-study comparison. Clin Pharmacol Drug Dev. 2014 Sep;3(5):406-16. doi: 10.1002/cpdd.118. Epub 2014 May 23. PMID 27129014